CLINICAL TRIAL: NCT07126262
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Vosoritide in Infants and Young Children With Hypochondroplasia, Aged 0 to < 36 Months
Brief Title: A Study of Vosoritide Versus Placebo in Children With Hypochondroplasia Aged 0 to < 36 Months
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-212
Record Dates: First submitted 2025-07-29; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypochondroplasia
MeSH Terms: conditions — Hypochondroplasia | interventions — vosoritide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vosoritide injection with vial and syringe (Experimental): Subcutaneous injection of recommended dose of vosoritide based on weight-band dosing once daily.
  Interventions: Drug: Vosoritide
- Placebo injection with vial and syringe (Placebo Comparator): Subcutaneous injection of recommended dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vosoritide — The vosoritide dose administered will be based on the participant's weight and will follow the weight-band dosing regimen approved for ACH
  Arms: Vosoritide injection with vial and syringe
Drug: Placebo — Subcutaneous injection of recommended dose of placebo
  Arms: Placebo injection with vial and syringe

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of daily administration of vosoritide in participants with HCH aged 0 to < 36 months over a 52-week period.

DETAILED DESCRIPTION:
Study 111-212 is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to assess the safety and efficacy of vosoritide versus placebo in infants and young children with HCH.

Eligible participants with documented HCH confirmed by genetic testing will be randomized in a 1:1 ratio to receive vosoritide or placebo. Participants will receive study treatment daily for 52 weeks by subcutaneous (SC) injection, followed by a 2-week safety follow-up visit. Vosoritide dosing will follow a weight-band regimen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must be 0 to < 36 months of age at randomization.
2. Participants must have a confirmed genetic diagnosis of HCH (obtained via whole genome sequencing; presence of a FGFR3 pathogenic variant associated with HCH).
3. Participants aged 0 to < 12 months must have a height Z-score of ≤ -1.0 SDS andparticipants aged ≥ 12 to < 36 months must have a height Z-score of ≤ -2.0 SDS in reference to the average stature of the same sex and age, as calculated using the Center for Disease Control and Prevention (CDC) growth charts.
4. Participant's weight at the Day 1 visit (pre-treatment) must be ≥ 3 kg.

Key Exclusion Criteria:

1. Short stature condition other than HCH (eg, ACH, trisomy 21, pseudoachondroplasia).
2. Have an unstable medical condition likely to require surgical intervention during the study period.
3. Taking any of the prohibited medications.
4. Have been treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids in the 6 months prior to Screening, or long-term treatment (> 3 months) at any time.
5. Require any investigational agent prior to completion of study period.
6. Have received another investigational product or investigational medical device within 30 days prior to the Screening visit.
7. Have used any other investigational product or investigational medical device for the treatment of HCH or short stature at any time.
8. Have current malignancy, history of malignancy, or currently under work-up for suspected malignancy.
9. Have known hypersensitivity to vosoritide or its excipients.
10. Have a condition or circumstance that, in the view of the investigator, places the participant at high risk for poor treatment compliance or for not completing the study.
11. Have any concurrent disease or condition that, in the view of the investigator, will interfere with study participation or safety evaluations, for any reason.

Ages: 0 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From baseline to end of treatment at 52 weeks
Incidence of serious adverse events versus placebo over the course of the study | From baseline to end of treatment at 52 weeks
Changes from baseline in standard clinical laboratory values (hematology, urinalysis, and chemistry) | At week 26, at week 52
Changes from baseline in heart rate | At week 13, at week 26, at week 39, at week 52
  Units of measure: bpm
Change from baseline in height Z-score | At week 52
Changes from baseline in respiratory rate | At week 13, at week 26, at week 39, at week 52
  Units of measure: breaths/min
Changes from baseline in temperature | At week 13, at week 26, at week 39, at week 52
  Units of measure: celsius
Changes from baseline in blood pressure | At week 13, at week 26, at week 39, at week 52
  Units of measure: mmHg

SECONDARY OUTCOMES:
Change in height | At week 52
Cumulative annualized growth velocity (AGV) | At week 52
6-month interval AGV | At week 26, at week 52
Change from baseline in upper to lower body segment ratio | At week 52
Change from baseline in arm span | At week 52
Change from baseline in total body (less head) bone mineral density (BMD) Z-score | At week 52
Change from baseline in lumbar spine BMD Z-score | At week 52
Change from baseline in total body (less head) bone mineral content (BMC) as measured by DXA | At week 52
Change from baseline in lumbar spine BMC as measured by DXA | At week 52
Area under the plasma vosoritide concentration time-curve from time 0 to infinity (AUC0-∞) | At week 26, at week 52
Area under the plasma vosoritide concentration time-curve from time 0 to the last measurable concentration (AUC0-t) | At week 26, at week 52
Elimination half-life of vosoritide (t½) | At week 26, at week 52
Apparent clearance of vosoritide | At week 26, at week 52
Apparent volume of distribution of vosoritide based upon the terminal phase (Vz/F) | At week 26, at week 52
Time vosoritide is present at maximum concentration (Tmax) | At week 26, at week 52
Maximum concentration (Cmax) of vosoritide in plasma | At week 26, at week 52
Change from pre-dose at pre-specified timepoints versus placebo in cyclic guanine monophosphate (cGMP) | At week 26 and week 52
Incidence of otitis media | From baseline to end of treatment at 52 weeks
Seizure frequency over the course of the study | From baseline to end of treatment at 52 weeks

CONTACTS AND LOCATIONS:
Locations (19):
- United States (9):
  - Phoenix Children's Hospital - Thomas Campus (Main), Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Benioff Children's Hospital - Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Minneasota Masonic Children's Hospital, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Children's Wisconsin - Fox Valley Hospital, Neenah, Wisconsin
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- France (2):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Paris
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron, Rhone-Alps
- Germany (3):
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätskinderklinik Magdeburg, Magdeburg, Saxony-Anhalt
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Rome
  - IRCCS Istituto Giannina Gaslini, Genova
- United Kingdom (2):
  - Myriad Trials, London, England
  - Great Ormond Street Hospital, London, England

IPD SHARING:
Plan to Share IPD: No